CLINICAL TRIAL: NCT00881881
Title: Clinical and Therapeutic Management of the Rheumatoid Arthritis in Spain
Brief Title: Study Evaluating the Clinical and Therapeutic Management of Rheumatoid Arthritis in Spain
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 0881A-102388
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with early RA

SUMMARY:
This is an epidemiological, multicenter, retrospective study to analyze the management of rheumatoid arthritis (RA) in usual clinical practice in Spain. Two groups of patients will be analyzed: individuals who have had RA for two years or less (the "early RA" group) and individuals who have had RA for more than 2 years and who currently meet the ACR criteria for RA (the "established RA" group).

ELIGIBILITY:
Inclusion criteria:

* Group 1: early RA : patients with disease lasting 2 years or less, considered by the investigator as an early RA
* Group 2: established RA: patients with disease lasting more than 2 years who meet the ACR criteria for RA

Exclusion criteria:

* Patients with any rheumatic disease different from RA
* Participation in any clinical trial or study in the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early RA and established RA treated in Rheumatology units in a real-world setting
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2006-12; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Therapeutic management of the RA (actual and 12 month follow-up) in a real-world setting. Descriptive analysis of sociodemographics and clinical variables for patients and sorted by group (early and established RA) for the last 12 months | 12 months

SECONDARY OUTCOMES:
Measurements of diagnostic and outcomes used in the common clinical practice. Degree of follow-up of the actual Spanish consensus on clinical and therapeutic management of patients with RA | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer